CLINICAL TRIAL: NCT02479230
Title: Pilot Trial of Type I-Polarized Autologous Dendritic Cell Vaccine Incorporating Tumor Blood Vessel Antigen-Derived Peptides in Patients With Metastatic Breast Cancer
Brief Title: Type I-Polarized Autologous Dendritic Cell Vaccine With Tumor Blood Vessel Antigen-Derived Peptides in Metastatic Breast Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joseph Baar, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Joseph Baar, MD, PhD, Associate Professor, Medicine, CWRU School of Medicine, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE3113; NCI-2014-00265 (Registry Identifier: CTRP)
Record Dates: First submitted 2015-06-19; First posted 2015-06-24 (Estimated); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer; Metastatic Breast Cancer
Keywords: vaccine; breast cancer; metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- vaccine: gemcitabine hydrochloride (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for 3 courses. Beginning 3, 7, or 10 days later, patients receive tumor blood vessel antigen peptide-pulsed alpha-type-1 polarized dendritic cell vaccine ID followed by a second vaccination 7 days later. Courses may repeat after at least 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: tumor blood vessel antigen peptide-pulsed alpha-type-1 polarized dendritic cell vaccine; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Biological: tumor blood vessel antigen peptide-pulsed alpha-type-1 polarized dendritic cell vaccine — Given ID
  Other Names: αDC1-TBVA vaccine
Drug: gemcitabine hydrochloride — Given IV
  Other Names: 1-(2-oxo-4-amino-1,2-dihydropyrimidin-1-yl)-2-deoxy-2,; 2-difluororibose hydrochloride,; 103882-84-4, 2'-deoxy-2',; 2'-difluorocytidine hydrochloride,; 2'deoxy-2',; 47762,; 613327,; dFdC,; dFdCyd,; difluorodeoxycytidine hydrochloride,; gemcitabine,; Gemzar,; LY-188011

SUMMARY:
This pilot clinical trial studies the safety of a dendritic cell vaccine when given with gemcitabine hydrochloride in treating patients with breast cancer that has spread beyond the breast and local lymph nodes to other organs in the body. The vaccine is made up of natural cells found in the blood, called dendritic cells, and peptides, or small fragments of protein which are loaded onto the dendritic cells. This combination may help activate the immune system against stromal cells, which are cells that help cancer cells survive in the body. Gemcitabine hydrochloride is a chemotherapy drug that is given before the vaccine to help shrink the tumor and control cells that may interfere with the activity of the vaccine. Interfering with the stromal cells that help support the growth of cancer cells may lead to the death of the cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety of gemcitabine hydrochloride (GEM) + alpha-type-1 dendritic cell (αDC1)-tumor blood vessel antigen (TBVA) vaccination (tumor blood vessel antigen peptide-pulsed alpha-type-1 polarized dendritic cell vaccine).

II. Assess the clinical response of metastatic breast cancer (MBC) to GEM + αDC1-TBVA vaccination.

III. Determine the clinical efficacy of GEM + αDC1-TBVA vaccination in generating T-helper 1 cell (Tc1) immunity.

IV. Correlate changes in myeloid-derived suppressor cells (MDSC) and regulatory T cells (Tregs) with the generation of anti-TBVA T-cell immunity.

OUTLINE:

Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1 and 8. Treatment repeats every 21 days for 3 courses. Beginning 3, 7, or 10 days later, patients receive tumor blood vessel antigen peptide-pulsed alpha-type-1 polarized dendritic cell vaccine intradermally (ID) followed by a second vaccination 7 days later. Courses may repeat after at least 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be human leukocyte antigen (HLA)-A2+
* Histologically confirmed breast cancer
* Patients must have evidence of metastatic disease measurable by Response Evaluation Criteria in Solid Tumors (RECIST) criteria or non-measurable lytic or mixed (lytic + blastic) bone lesions in the absence of measurable disease; Note: Measurable lesions include lytic or mixed (lytic + blastic) bone lesions, with an identifiable 10 mm soft tissue component that meets the measurability criteria per RECIST
* There is no limit to the number of prior systemic treatment regimens
* Patients must have a life expectancy of > 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Prior GEM therapy is acceptable as long as the last dose was ≥ 3 months from registration on this study
* Patients may have treated and stable brain metastases; they must be off steroids and must have had stable brain metastases for at least 6 months
* White blood cell (WBC) > 3.0 x 10^9/L
* Platelets > 100 x 10^9/L
* Hemoglobin (Hgb) ≥ 10.0 gm/dl
* Creatinine < 1.5 mg/dl
* Bilirubin (total) < 2.0 ml/dl
* Aspartate aminotransferase (AST) < 5.0 x normal institutional limits
* Alkaline phosphatase < 2.5 upper limit of normal (ULN) (< 10 x ULN in presence of bone metastases)
* Serum calcium ≤ 12 mg/dl
* International normalized ratio (INR) < 1.5, except for subjects receiving warfarin therapy; for subjects who are receiving warfarin for prophylaxis or treatment of thrombosis, INR values should be carefully monitored while patients are on study
* All patients must be informed of the investigational nature of this study and must provide written informed consent in accordance with institutional and federal guidelines; a copy of the informed consent document signed by the patient must be given to the patient
* Patients must have a negative pregnancy test by urinalysis
* Use of an effective means of contraception (men and women) is mandated in subjects of child-bearing potential; female subjects will be advised that they not become pregnant for at least one month after completing participation in the study; avoiding sexual activity is the only certain method to prevent pregnancy; however, if subjects choose to be sexually active, they should use an appropriate "double barrier" method of birth control (such as female use of a diaphragm, intrauterine device [IUD], or contraceptive sponge, in addition to male use of a condom) or the use of prescribed "birth control" pills, injections, or implants

Exclusion Criteria:

* HLA-A2 negative patients
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness
* Presence of bleeding diathesis
* Current treatment on another clinical trial
* Patients with organ allografts
* Pregnancy or breast-feeding; female patients must be surgically sterile or be post-menopausal, or must agree to use effective contraception during the period of therapy; all female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment; male patients must be surgically sterile or must agree to use effective contraception during the period of therapy; the definition of effective contraception will be based on the judgment of the principal investigator or a designated associate
* Other severe acute or chronic medical or psychiatric conditions, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-07-17 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Number of toxicities | 30 days after completion of study
  Incidence of toxicities, evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0

SECONDARY OUTCOMES:
mean change in Type-1 immune function | 24 weeks after treatment
  Average immune response as measured by the interferon gamma [IFN-γ] cluster of differentiation (CD)8+ T cell (Tc1) response to the vaccine-associated TBVA peptides.
Number of patients with clinical response | Up to 30 days after study is complete
  Clinical response as assessed using RECIST criteria.

OTHER OUTCOMES:
Change in Treg levels | 24 weeks after treatment
  The correlation between vaccine-induced anti-TBVA T-cell immunity and changes in Tregs and MDSC levels will be estimated using Pearson correlation coefficient
Changes in MDSC levels | 24 weeks after treatment
  The correlation between vaccine-induced anti-TBVA T-cell immunity and changes in Tregs and MDSC levels will be estimated using Pearson correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Baar, MD, PhD, Principal Investigator — Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania